CLINICAL TRIAL: NCT03656705
Title: Clinical Investigation of Chimeric Costimulatory Converting Receptor(CCCR)-Modified NK92 Cells in Previously Treated Advanced Non-small Cell Lung Carcinoma
Brief Title: CCCR-NK92 Cells Immunotherapy for Non-small Cell Lung Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Henan Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNK-101
Record Dates: First submitted 2018-07-11; First posted 2018-09-04 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CCCR-NK92 cells immunotherapy (Experimental): Preparation of CCCR-NK92 cells suspended in a saline and plasma solution.
  Interventions: Biological: CCCR-NK92 cells

INTERVENTIONS:
Biological: CCCR-NK92 cells — CCCR-NK92 cells will be administered intravenously over 1h. The starting dose of CCCR-NK92 cells will be 1×10e7-1×10e8,twice a week. The first evaluation of the efficacy after 3 weeks of treatment.

SUMMARY:
The purpose of this clinical investigation is to evaluate the safety and effects of CCCR-modified NK92(CCCR-NK92)infusions in previously treated advanced non-small cell lung carcinoma(NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* 1.Male and female subjects with non-small cell lung carcinoma in patients with no available curative treatment options who have limited prognosis(≧3 months)with currently available therapies will be enrolled.
* 2.The last cytotoxic drug, radiotherapy or surgery≧4 weeks.
* 3.HB≧90g/L, ANC≧1.5×10e9/L, PLT≧80×10e9/L, TBIL≦1.5×upper limit of nomal, ALT/AST≦2.5×upper limit of nomal, ALT/AST≦5×upper limit of nomal if have liver metastasis, Cr≦1.5×upper limit of nomal or CCr≧60ml/min.

Exclusion Criteria:

* 1.Pregnancy or breastfeeding.
* 2.Known HIV, HBV or HCV infection.
* 3.Active antoimmune disease.
* 4.History of severe immediate hypersensitivity to any of the biological products including penicillin.
* 5.Severe psychiatric disorder which might interfere with the study treatment or examination.
* 6.Chronic heart failure NYHA≧III.
* 7.Simultaneous participation in another clinical trial within 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-09-29 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events evaluated with CTCAE,version 4.0 | 3 months
  Safety evaluation
Objective Response Rate | up to one year
  Non-small cell lung carcinoma to CCCR-NK92 cell infusions

SECONDARY OUTCOMES:
Disease Control Rate | up to one year
Progression-free Survival | up to one year
Overall Survival | up to one year

CONTACTS AND LOCATIONS:
Locations (1):
- The first Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan, China

IPD SHARING:
Plan to Share IPD: No